CLINICAL TRIAL: NCT04934111
Title: A Clinical Trial to Assess the Safety and Immunogenicity of LNP-nCOV saRNA-02, a Self-amplifying Ribonucleic Acid (saRNA) Vaccine, in SARS-CoV-2 Seronegative and Seropositive Uganda Population
Brief Title: Safety and Immunogenicity of LNP-nCOV saRNA-02 Vaccine Against SARS-CoV-2, the Causative Agent of COVID-19
Acronym: COVAC-Uganda
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: COVAC Uganda
Record Dates: First submitted 2021-06-10; First posted 2021-06-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: SARS-CoV-2, LNP-nCOV saRNA-02, COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This phase I clinical study builds on clinical experience using the LNP nCoV saRNA vaccine currently under evaluation in COVAC1 (Being conducted in the UK). The trial will be conducted in 18-45 year olds in a single centre supervised by the Chief Investigator, by allocating the 42 participants into two groups, based on seroconversion status. These will include 21 SARS-CoV-2 seronegative and 21 SARs-CoV-2 seropositive individuals. Participants in each group will be given a dose of 5.0ug at 0 weeks and 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LNP-nCOV saRNA-02 Vaccine arm (Experimental): Participants that have evidence of previous infection with SARS-CoV-2 and those with no evidence of previous infection will all receive receive LNP-nCOV saRNA-02 Vaccine. Both groups will be given a dose of 5.0ug at 0 weeks and 4 weeks.
  Interventions: Drug: LNP-nCOV saRNA-02 Vaccine

INTERVENTIONS:
Drug: LNP-nCOV saRNA-02 Vaccine — a self-amplifying ribonucleic acid (saRNA) vaccine encoding the S glycoprotein of SARS-CoV-2, the causative agent of COVID-19

SUMMARY:
COVAC Uganda is a study that is looking at the use of an innovative self-amplifying RNA (saRNA) vaccine (LNP-nCOV saRNA-02) against the virus (SARS-CoV-2) that causes COVID-19 and assessing the immune response in SARS-CoV-2 antibody seronegative and seropositive individuals. saRNA is designed to amplify the quantity of RNA upon injection to produce further antigen, thereby enabling lower doses for administration. In the trial "COVAC1", Imperial College London is currently evaluating one COVID-19 saRNA vaccine candidate in doses from 0.1-10ug for individuals who are seronegative for SARS-CoV-2 antibodies at baseline. Interim analyses of COVAC1 has shown a dose dependent response; however, up to 50% of seronegative participants receiving doses of 2.5-10ug do not seroconvert. The investigators hypothesize that a lack of seroconversion is due to type I and III interferon (IFN) production, which can inhibit translation and degrade cellular mRNA. Another variable that can enhance antibody production is serological history: recent studies have shown that seropositive individuals respond significantly better than naïve individuals who received the Pfizer or Moderna RNA-based COVID-19 vaccine. Therefore, designing the saRNA backbone to dampen IFN production and evaluating this in individuals seropositive at baseline will inform the optimised use of this innovative technology. In COVAC Uganda, the investigators aim to test an saRNA vaccine modified to dampen the activation of type I and III IFN, to increase antibody production, for individuals who are seronegative and seropositive for SARS-CoV-2 antibodies at baseline, to evaluate whether people with pre-existing seropositivity have enhanced immune responses compared to those without. This trial is NOT looking at whether or not the vaccine is effective in terms of protection. It is just assessing whether and how well the immune system responds based on SARS-CoV-2 antibodies at baseline and its safety.

DETAILED DESCRIPTION:
Background The ongoing pandemic coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) emerged in humans in China sometime between October to November 2019, and the disease coronavirus infectious disease 2019 (COVID-19) was identified in China in December 2019.

By the end of January 2021, SARS-CoV-2 had infected with confirmed diagnosis over 106 million people worldwide, resulting in over 2.3 million deaths and over 59 million people recovered from infection. This yields a nominal infection fatality rate (IFR) of ~2%, and around 10% of infected people have been left with health effects lasting for 6 months or more. As of 8 March 2021, Uganda had reported 40,452 coronavirus cases and 334 deaths. Through COVAX, Uganda started rolling out the AstraZeneca vaccine (adenoviral based) from 10 March 2021.

The developing assessment is that the only way the world can exit from the COVID-19 pandemic is through the deployment of an effective vaccine. A number of vaccines have been developed and received emergency use authorization by the United States Food and Drug Administration and/or the World Health Organization. Examples include Pfizer-BioNTech and Moderna's messenger ribonucleic acid (mRNA)-based vaccines which have both shown efficacy at 95%; Oxford-AstraZeneca's ChAdOx1 nCoV-19 and Johnson and Johnson's adenovirus based vaccines which have demonstrated efficacies of 70% and 66% respectively. The problem comes with the scale needed and the time frame in which vaccines need to be developed and deployed. A self-amplifying RNA (saRNA) vaccine provides a novel, feasible, and time-sensitive solution to contribute to addressing the SARS-CoV-2 problem, either during the current pandemic or for ongoing seasonal epidemics.

Studies have demonstrated that nucleic acid-based vaccination can protect against viral infections in non-human primate (NHP) studies, providing proof of concept that gene-based vaccination can induce protective antibodies. However, DNA vaccines require multiple immunizations with the use of electroporation to induce significant immune responses in humans. Non-replicating mRNA-based therapeutics typically require high doses of RNA (100-600 µg). The requirement for high doses, and associated cost, suggest non-replicating mRNA may struggle to produce the potential hundreds of millions of doses required to rapidly respond to a pandemic. In contrast, small animal and non-human primate (NHP) experiments suggest that saRNA induces significantly enhanced responses in comparison to either DNA vaccines delivered with electroporation or mRNA. Indeed, a single immunization with a saRNA vaccine has shown protection against Ebola virus in animal models. Should a ≤10 µg dose of saRNA provide protection from COVID-19, this would provide critical advantages for manufacturing where 100,000 doses can by synthesized in a one liter reaction volume. In contrast to viral vectors, lack of anti-vector immunity provides the opportunity for repeat immunizations with multiple RNA-encoded immunogens.

The first generation saRNA vaccine (LNP-nCoV-saRNA) is already undergoing safety assessment in humans in the COVAC1 trial in the United Kingdom. The safety of this first generation saRNA vaccine has been assessed initially in healthy young adults i.e., 15 participants aged 18-45 years, given one of three different doses (0.1, 0.3 and 1 µg) by injection into the muscle, going slowly from the lowest to the highest over a period of several weeks. To date, there have been no reported serious adverse events (SAEs) associated with this vaccine and a low frequency of Grade 2 events. An additional 35 volunteers have been randomized across each dose. To date, 105 healthy subjects have received two immunizations across each dose, with few Grade 2 events. All participants have safely received both doses. Initial assessment of the first 15 subjects indicates that although the vaccine shows a good safety profile, the levels of seroconversion (75% for the 1ug dose) and binding antibody are lower than anticipated from preclinical models. Indeed, data generated to date suggest responses are at the lower end of a dose response curve. An additional expansion phase has been initiated to explore three higher doses 2.5, 5 and 10ug. The disconnect between human immune response to the vaccine and preclinical models suggests that the level of saRNA expression in humans is less effective than in small animal models. Current data indicate that 5ug dose administered at 0 and 4 weeks induces an acceptable immune response to most (83%) individuals 4-weeks post 2nd vaccination.

The investigators have improved on this initial design (COVAC1) with the modified vector, LNP-nCOV saRNA-02, which is to be investigated within this clinical trial.

This study (COVAC Uganda) will evaluate an innovative saRNA vaccine (LNP-nCOV saRNA-02) designed to increase vaccine potency by shielding the saRNA from cellular proteins known to reduce saRNA expression. The investigators anticipate the safety profile of the modified vaccine to be highly similar to the first generation vaccine already undergoing human trials. COVAC Uganda will use the same assessment criteria as the COVAC1 study designed to see how well the immune system has been activated using different dose levels of the modified vaccine. COVAC Uganda will also enrol SARS-CoV-2 seropositive individuals to evaluate the immune response based on serological history. Seronegative and seropositive participants aged 18-45 will be given one dose of 5.0 ug at 0 weeks and 4 weeks. Seronegative is defined as IgG ≤ 10 AU mL-1 or IgM ≤ 10 AU mL-1, and seropositive is defined as IgG ≥ 10 AU mL-1 or IgM ≥ 10 AU mL-1. The vaccine is given by injection into the muscle of the upper arm. There are likely to be mild side-effects near to the injection site. As observed in COVAC1, there may also be more general side-effects such as headache, temperature and chills. Participants will be asked to record any symptoms in a vaccine diary. In order to see how well the immune system is responding, participants will need to give blood samples several times during the first 6 weeks; then monthly for a few months; then at 6 months.

The investigators predict that the modified vaccine will induce higher levels of neutralising antibodies than the first generation saRNA vaccine. However, if any of the doses do not induce an adequate immune response, there is no known reason why participants who received those doses could not be offered a further booster immunisation with LNP-nCOV saRNA-02 at a dose that has been shown to be safe. Also there is no known reason why participants in COVAC Uganda could not be immunised with other approved SARS-CoV-2 vaccines, including vectored or adjuvanted vaccines, should they be shown to be safe and effective.

Study Rationale This SARS-CoV-2 pandemic has infected over 106 million people and killed over 2.3 million people. As a novel zoonotic virus, no herd immunity is present and the only widely available interventions to date are social distancing to reduce pressure on intensive care beds and health systems, but this is not sustainable for economic reasons. Clinical trials of antivirals and other drug therapies are ongoing but the intervention most likely to mitigate the long-term medical, social and economic impact of the pandemic remains population-wide immunisation.

Despite successfully approved COVID-19 vaccines being rolled out, substantially more candidates are needed to supply 4.265 billion doses for the world's healthcare workers, adults >65 age, and people at higher risk (with co-morbidities such as diabetes, cardiovascular disease, cancer, obesity or chronic respiratory disease), let alone doses for younger or healthier cohorts.

Recent evidence suggests that immune responses to messenger RNA vaccines is enhanced for individuals previously infected by SARS-CoV-2. This trial investigates the role of seroconversion on the impact of a self-amplifying RNA vaccine candidate, and it will inform on the possible application of LNP-nCOV saRNA-02 as a COVID-19 booster candidate for previously infected individuals.

Pre-clinical data suggest that the LNP-nCOV saRNA-02 vaccine encoding a prefusion stabilised version of the S-glycoprotein will elicit neutralising antibodies in a higher proportion of individuals than natural infection (<50%), and that the LNP-nCOV saRNA-02 vaccine may provide increased immunogenicity and/or dose reduction over the first generation construct as well as for seropositive individuals.

Study Design This is a phase I clinical study which will build on clinical experience using the LNP nCoV saRNA vaccine currently under evaluation in COVAC1 in the UK. The trial will be conducted in 18-45 year olds in a single centre supervised by the Chief/principal Investigator, by allocating 42 participants into two groups, based on seroconversion status.

Subject Population The study will be conducted in healthy young adults as these individuals generate the most robust responses (18-45 years). Both male and female participants will be included and the trial site will attempt to keep an equal proportion, although the priority will be to ensure timely accrual to the trial.

Dosage and Admiration

Participants will each receive one IM dose of 5 ug of LNP-nCOV saRNA-02, into the deltoid muscle at Week 0 and Week 4 as indicated in the table below:

Study component Serological Status Route Dose Vaccination 1 Vaccination 2 Serological Group SARS-CoV-2 negative antibodies IM 5.0 ug LNP-CoV mod-saRNA-02 Week 0

Visit 2 Week 4

Visit 5 SARS-CoV-2 positive antibodies IM 5.0 ug LNP-CoV mod-saRNA-02 Week 0

Visit 2 Week 4

Visit 5

Safety Evaluations Vaccines are associated with a number of well-characterized local, systemic and laboratory reactions referred to as solicited adverse events. These adverse events will be purposively collected.

Local and systemic assessments will take place on the day of each injection before the injection, and 60 minutes after the injection. Participants should remain at the clinic for at least one hour after each injection.

Participants will be provided with Vaccine diary cards to assist collection and grading of adverse events that start within 7 days of the injection. Study staff will go through the list of solicited adverse events in a structured interview and record these together with grade on the appropriate eCRF in the REDCap database. If any of the events reported at one of the phone visits are moderately severe (grade 2) or worse, participants will be invited to the clinic for review.

Blood (~10 mL) for routine safety parameters will be collected at all study visits. If the total bilirubin is elevated, study staff will request a result for conjugated bilirubin in order to grade the abnormality and determine any action to be taken with respect to further investigation and interruption to the vaccine schedule.

Vital signs (BP, HR, oxygen saturation and oral temperature) will be measured at every study visit.

Physical examinations of the injection site, and other body systems if indicated, will be performed on the day of each vaccination, and 1 week after. Symptom-directed physical examinations will be performed at all other follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults from the following aged 18-45 years on the day of screening
2. At similar risk of acquiring SARS-CoV-2 infection to the general population
3. Willing and able to provide informed consent
4. If female and of childbearing potential, willing to use a highly effective method of contraception from screening until 18 weeks after last injection
5. If male and not sterilised, willing to avoid impregnating female partners from screening until 18 weeks after last injection
6. Willing to avoid all other vaccines from within 4 weeks before the first injection through to 22 weeks after the second injection
7. Willing and able to comply with visit schedule, complete vaccine diaries and provide samples
8. Willing to grant authorised persons access to his/her trial-related medical record and GP records either directly or indirectly

Exclusion Criteria:

1. Pregnant or lactating
2. Has a significant clinical history, physical finding on clinical examination during screening, or presence of a disease that is active or requires treatment to control it, including cardiac, respiratory, endocrine, metabolic, autoimmune, liver, neurological, oncological, psychiatric, immunosuppressive/immunodeficient or other disorders which in the opinion of the investigator is not compatible with healthy status, increases the risk of severe COVID-19, may compromise the volunteer's safety, preclude vaccination or compromise interpretation of the immune response to vaccine. Individuals with mild/moderate, well-controlled comorbidities are allowed.
3. History of anaphylaxis or angioedema
4. Active SARS-CoV-2 infection at enrolment, based on DNA-PCR testing
5. Discordant RDT result
6. History of severe or multiple allergies to drugs or pharmaceutical agents
7. History of severe local or general reaction to vaccination defined as:

   1. local: extensive, indurated redness and swelling involving most of the arm, not resolving within 72 hours
   2. general: fever ≥39.5 °C within 48 hours; bronchospasm; laryngeal edema; collapse; convulsions or encephalopathy within 72 hours
8. Ever received an experimental vaccine against COVID-19
9. Receipt of any immunosuppressive agents within 18 weeks of screening by any route other than topical
10. Detection of antibodies to hepatitis C
11. Detection of antibodies to HIV
12. Grade 1 and above abnormalities in routine laboratory parameters using the FDA toxicity table Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. https://www.fda.gov/media/73679/download
13. Participating in another clinical trial with an investigational drug or device, or treated with an investigational drug within 28 days of screening.
14. Has received an immunisation within 28 days of screening
15. Has received an authorised COVID-19 vaccine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with solicited local injection site reactions | 7 days after each injection
  Number of participants with solicited local injection site reactions starting within 7 days of administration of the vaccine: pain, tenderness, erythema, swelling
Number of participants with solicited systemic reactions starting within 7 days of administration of the vaccine | 7 days after each injection
  Number of participants with solicited systemic reactions starting within 7 days of administration of the vaccine: pyrexia, fatigue, myalgia, headache, chills, arthralgia
Number of participants with unsolicited adverse reactions (ARs) throughout the study | 6 months
  Number of participants with unsolicited adverse reactions (ARs) throughout the study period (including serious ARs)
Number of participants with serious Adverse Events | 6 months
  Number of participants with serious Adverse Events
Number of participants with unsolicited adverse events | 6 months
  Number of participants with unsolicited adverse events throughout the study period
The titer of serum neutralizing antibodies 2 weeks after the second vaccination in the SARS-CoV-2 pseudovirus-based neutralization assay | from day 1, through six months
  The titer of serum neutralizing antibodies 2 weeks after the second vaccination in the SARS-CoV-2 pseudovirus-based neutralization assay
The titer of vaccine-induced serum IgG binding antibody responses to the SARS-CoV-2 S glycoprotein 2 weeks after the first and second vaccinations | from day 1, through six months
  The titer of vaccine-induced serum IgG binding antibody responses to the SARS-CoV-2 S glycoprotein 2 weeks after the first and second vaccinations

SECONDARY OUTCOMES:
Cell-mediated vaccine-induced immune responses measured by T- and B- cell ELISpot in study participants | from day 1, through six months
  Cell-mediated vaccine-induced immune responses measured by T- and B- cell ELISpot in study participants
Cell-mediated vaccine-induced immune responses measured by flow cytometry and intracellular cytokine staining in study participants | from day 1, through six months
  Cell-mediated vaccine-induced immune responses measured by flow cytometry and intracellular cytokine staining in study participants
The profile of class and sub-class of antibody response | from day 1, through six months
  The profile of class and sub-class of antibody response
Laboratory markers of infection and infection-induced immunity | through the 6 months of the trial
  Laboratory markers of infection and infection-induced immunity
Incidence of thrombocytopenia of any grade confirmed on repeat testing if possible | Through 6 months of the trial
  Incidence of thrombocytopenia of any grade confirmed on repeat testing if possible

CONTACTS AND LOCATIONS:
Overall Officials: Pontiano Kaleebu, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- MRC/UVRI & LSHTM Uganda Research Unit, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to the Imperial College London data sharing policies, adherent to General Data Protection Regulations (https://www.imperial.ac.uk/research-and-innovation/research-office/research-governance-and-integrity/what-is-research-governance-and-integrity/data-protection---information-for-participants/) and the MRC/UVRI & LSHTM Uganda Research Unit Data Sharing Policy (https://www.mrcuganda.org/publications/data-sharing-policy) and controlled access approach.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available for sharing after study completion. Data may be assumed to be indefinitely available after that point until otherwise stated.
Access Criteria: Criteria may be accessed through link below
URL: https://www.imperial.ac.uk/research-and-innovation/research-office/research-governance-and-integrity/what-is-research-governance/data-protection---information-for-participants/

REFERENCES:
- [Background] Herbert AS, Kuehne AI, Barth JF, Ortiz RA, Nichols DK, Zak SE, Stonier SW, Muhammad MA, Bakken RR, Prugar LI, Olinger GG, Groebner JL, Lee JS, Pratt WD, Custer M, Kamrud KI, Smith JF, Hart MK, Dye JM. Venezuelan equine encephalitis virus replicon particle vaccine protects nonhuman primates from intramuscular and aerosol challenge with ebolavirus. J Virol. 2013 May;87(9):4952-64. doi: 10.1128/JVI.03361-12. Epub 2013 Feb 13. PMID 23408633
- [Background] Li W, Ye L, Carrion R Jr, Mohan GS, Nunneley J, Staples H, Ticer A, Patterson JL, Compans RW, Yang C. Characterization of Immune Responses Induced by Ebola Virus Glycoprotein (GP) and Truncated GP Isoform DNA Vaccines and Protection Against Lethal Ebola Virus Challenge in Mice. J Infect Dis. 2015 Oct 1;212 Suppl 2(Suppl 2):S398-403. doi: 10.1093/infdis/jiv186. Epub 2015 Apr 14. PMID 25877553
- [Background] Cashman KA, Broderick KE, Wilkinson ER, Shaia CI, Bell TM, Shurtleff AC, Spik KW, Badger CV, Guttieri MC, Sardesai NY, Schmaljohn CS. Enhanced Efficacy of a Codon-Optimized DNA Vaccine Encoding the Glycoprotein Precursor Gene of Lassa Virus in a Guinea Pig Disease Model When Delivered by Dermal Electroporation. Vaccines (Basel). 2013 Jul 18;1(3):262-77. doi: 10.3390/vaccines1030262. PMID 26344112
- [Background] Grant-Klein RJ, Altamura LA, Badger CV, Bounds CE, Van Deusen NM, Kwilas SA, Vu HA, Warfield KL, Hooper JW, Hannaman D, Dupuy LC, Schmaljohn CS. Codon-optimized filovirus DNA vaccines delivered by intramuscular electroporation protect cynomolgus macaques from lethal Ebola and Marburg virus challenges. Hum Vaccin Immunother. 2015;11(8):1991-2004. doi: 10.1080/21645515.2015.1039757. PMID 25996997
- [Background] Shedlock DJ, Aviles J, Talbott KT, Wong G, Wu SJ, Villarreal DO, Myles DJ, Croyle MA, Yan J, Kobinger GP, Weiner DB. Induction of broad cytotoxic T cells by protective DNA vaccination against Marburg and Ebola. Mol Ther. 2013 Jul;21(7):1432-44. doi: 10.1038/mt.2013.61. Epub 2013 May 14. PMID 23670573
- [Background] Grant-Klein RJ, Van Deusen NM, Badger CV, Hannaman D, Dupuy LC, Schmaljohn CS. A multiagent filovirus DNA vaccine delivered by intramuscular electroporation completely protects mice from ebola and Marburg virus challenge. Hum Vaccin Immunother. 2012 Nov 1;8(11):1703-6. doi: 10.4161/hv.21873. Epub 2012 Aug 24. PMID 22922764
- [Background] Li L, Petrovsky N. Molecular mechanisms for enhanced DNA vaccine immunogenicity. Expert Rev Vaccines. 2016;15(3):313-29. doi: 10.1586/14760584.2016.1124762. Epub 2015 Dec 28. PMID 26707950
- [Background] Alberer M, Gnad-Vogt U, Hong HS, Mehr KT, Backert L, Finak G, Gottardo R, Bica MA, Garofano A, Koch SD, Fotin-Mleczek M, Hoerr I, Clemens R, von Sonnenburg F. Safety and immunogenicity of a mRNA rabies vaccine in healthy adults: an open-label, non-randomised, prospective, first-in-human phase 1 clinical trial. Lancet. 2017 Sep 23;390(10101):1511-1520. doi: 10.1016/S0140-6736(17)31665-3. Epub 2017 Jul 25. PMID 28754494
- [Background] Sahin U, Kariko K, Tureci O. mRNA-based therapeutics--developing a new class of drugs. Nat Rev Drug Discov. 2014 Oct;13(10):759-80. doi: 10.1038/nrd4278. Epub 2014 Sep 19. PMID 25233993
- [Background] Feldman RA, Fuhr R, Smolenov I, Mick Ribeiro A, Panther L, Watson M, Senn JJ, Smith M, Almarsson Ӧ, Pujar HS, Laska ME, Thompson J, Zaks T, Ciaramella G. mRNA vaccines against H10N8 and H7N9 influenza viruses of pandemic potential are immunogenic and well tolerated in healthy adults in phase 1 randomized clinical trials. Vaccine. 2019 May 31;37(25):3326-3334. doi: 10.1016/j.vaccine.2019.04.074. Epub 2019 May 10. PMID 31079849
- [Background] Kis Z, Shattock R, Shah N, Kontoravdi C. Emerging Technologies for Low-Cost, Rapid Vaccine Manufacture. Biotechnol J. 2019 Jan;14(1):e1800376. doi: 10.1002/biot.201800376. Epub 2018 Dec 10. Erratum In: Biotechnol J. 2019 Jul;14(7):1-2. doi: 10.1002/biot.201970055. PMID 30537361
- [Background] Wrapp D, Wang N, Corbett KS, Goldsmith JA, Hsieh CL, Abiona O, Graham BS, McLellan JS. Cryo-EM structure of the 2019-nCoV spike in the prefusion conformation. Science. 2020 Mar 13;367(6483):1260-1263. doi: 10.1126/science.abb2507. Epub 2020 Feb 19. PMID 32075877
- [Background] Ljungberg K, Liljestrom P. Self-replicating alphavirus RNA vaccines. Expert Rev Vaccines. 2015 Feb;14(2):177-94. doi: 10.1586/14760584.2015.965690. Epub 2014 Oct 1. PMID 25269775
- [Background] Ulmer JB, Mansoura MK, Geall AJ. Vaccines 'on demand': science fiction or a future reality. Expert Opin Drug Discov. 2015 Feb;10(2):101-6. doi: 10.1517/17460441.2015.996128. Epub 2015 Jan 13. PMID 25582273
- [Background] Brito LA, Kommareddy S, Maione D, Uematsu Y, Giovani C, Berlanda Scorza F, Otten GR, Yu D, Mandl CW, Mason PW, Dormitzer PR, Ulmer JB, Geall AJ. Self-amplifying mRNA vaccines. Adv Genet. 2015;89:179-233. doi: 10.1016/bs.adgen.2014.10.005. Epub 2014 Dec 4. PMID 25620012
- [Background] Erwin-Cohen RA, Porter AI, Pittman PR, Rossi CA, DaSilva L. Human transcriptome response to immunization with live-attenuated Venezuelan equine encephalitis virus vaccine (TC-83): Analysis of whole blood. Hum Vaccin Immunother. 2017 Jan 2;13(1):169-179. doi: 10.1080/21645515.2016.1227900. Epub 2016 Nov 21. PMID 27870591
- [Background] Bernstein DI, Reap EA, Katen K, Watson A, Smith K, Norberg P, Olmsted RA, Hoeper A, Morris J, Negri S, Maughan MF, Chulay JD. Randomized, double-blind, Phase 1 trial of an alphavirus replicon vaccine for cytomegalovirus in CMV seronegative adult volunteers. Vaccine. 2009 Dec 11;28(2):484-93. doi: 10.1016/j.vaccine.2009.09.135. Epub 2009 Oct 24. PMID 19857446
- [Background] Crank MC, Ruckwardt TJ, Chen M, Morabito KM, Phung E, Costner PJ, Holman LA, Hickman SP, Berkowitz NM, Gordon IJ, Yamshchikov GV, Gaudinski MR, Kumar A, Chang LA, Moin SM, Hill JP, DiPiazza AT, Schwartz RM, Kueltzo L, Cooper JW, Chen P, Stein JA, Carlton K, Gall JG, Nason MC, Kwong PD, Chen GL, Mascola JR, McLellan JS, Ledgerwood JE, Graham BS; VRC 317 Study Team. A proof of concept for structure-based vaccine design targeting RSV in humans. Science. 2019 Aug 2;365(6452):505-509. doi: 10.1126/science.aav9033. PMID 31371616
- [Background] Lui PY, Wong LR, Ho TH, Au SWN, Chan CP, Kok KH, Jin DY. PACT Facilitates RNA-Induced Activation of MDA5 by Promoting MDA5 Oligomerization. J Immunol. 2017 Sep 1;199(5):1846-1855. doi: 10.4049/jimmunol.1601493. Epub 2017 Jul 31. PMID 28760879
- [Background] Siu KL, Yeung ML, Kok KH, Yuen KS, Kew C, Lui PY, Chan CP, Tse H, Woo PC, Yuen KY, Jin DY. Middle east respiratory syndrome coronavirus 4a protein is a double-stranded RNA-binding protein that suppresses PACT-induced activation of RIG-I and MDA5 in the innate antiviral response. J Virol. 2014 May;88(9):4866-76. doi: 10.1128/JVI.03649-13. Epub 2014 Feb 12. PMID 24522921
- [Background] Batool M, Shah M, Patra MC, Yesudhas D, Choi S. Structural insights into the Middle East respiratory syndrome coronavirus 4a protein and its dsRNA binding mechanism. Sci Rep. 2017 Sep 12;7(1):11362. doi: 10.1038/s41598-017-11736-6. PMID 28900197
- [Background] Rabouw HH, Langereis MA, Knaap RC, Dalebout TJ, Canton J, Sola I, Enjuanes L, Bredenbeek PJ, Kikkert M, de Groot RJ, van Kuppeveld FJ. Middle East Respiratory Coronavirus Accessory Protein 4a Inhibits PKR-Mediated Antiviral Stress Responses. PLoS Pathog. 2016 Oct 26;12(10):e1005982. doi: 10.1371/journal.ppat.1005982. eCollection 2016 Oct. PMID 27783669
- [Background] McKay PF, Hu K, Blakney AK, Samnuan K, Brown JC, Penn R, Zhou J, Bouton CR, Rogers P, Polra K, Lin PJC, Barbosa C, Tam YK, Barclay WS, Shattock RJ. Self-amplifying RNA SARS-CoV-2 lipid nanoparticle vaccine candidate induces high neutralizing antibody titers in mice. Nat Commun. 2020 Jul 9;11(1):3523. doi: 10.1038/s41467-020-17409-9. PMID 32647131
- [Background] Slovin SF, Kehoe M, Durso R, Fernandez C, Olson W, Gao JP, Israel R, Scher HI, Morris S. A phase I dose escalation trial of vaccine replicon particles (VRP) expressing prostate-specific membrane antigen (PSMA) in subjects with prostate cancer. Vaccine. 2013 Jan 30;31(6):943-9. doi: 10.1016/j.vaccine.2012.11.096. Epub 2012 Dec 13. PMID 23246260
- [Background] Demoulins T, Milona P, Englezou PC, Ebensen T, Schulze K, Suter R, Pichon C, Midoux P, Guzman CA, Ruggli N, McCullough KC. Polyethylenimine-based polyplex delivery of self-replicating RNA vaccines. Nanomedicine. 2016 Apr;12(3):711-722. doi: 10.1016/j.nano.2015.11.001. Epub 2015 Dec 1. PMID 26592962
- [Background] Vogel AB, Lambert L, Kinnear E, Busse D, Erbar S, Reuter KC, Wicke L, Perkovic M, Beissert T, Haas H, Reece ST, Sahin U, Tregoning JS. Self-Amplifying RNA Vaccines Give Equivalent Protection against Influenza to mRNA Vaccines but at Much Lower Doses. Mol Ther. 2018 Feb 7;26(2):446-455. doi: 10.1016/j.ymthe.2017.11.017. Epub 2017 Dec 5. PMID 29275847
- [Background] Hoy SM. Patisiran: First Global Approval. Drugs. 2018 Oct;78(15):1625-1631. doi: 10.1007/s40265-018-0983-6. PMID 30251172
- [Background] NCT04283461. Safety and Immunogenicity Study of 2019-nCoV Vaccine (mRNA-1273) to Prevent SARS-CoV-2 Infection
- [Background] Lokugamage KG, Yoshikawa-Iwata N, Ito N, Watts DM, Wyde PR, Wang N, Newman P, Kent Tseng CT, Peters CJ, Makino S. Chimeric coronavirus-like particles carrying severe acute respiratory syndrome coronavirus (SCoV) S protein protect mice against challenge with SCoV. Vaccine. 2008 Feb 6;26(6):797-808. doi: 10.1016/j.vaccine.2007.11.092. Epub 2007 Dec 26. PMID 18191004
- [Background] Yasui F, Kai C, Kitabatake M, Inoue S, Yoneda M, Yokochi S, Kase R, Sekiguchi S, Morita K, Hishima T, Suzuki H, Karamatsu K, Yasutomi Y, Shida H, Kidokoro M, Mizuno K, Matsushima K, Kohara M. Prior immunization with severe acute respiratory syndrome (SARS)-associated coronavirus (SARS-CoV) nucleocapsid protein causes severe pneumonia in mice infected with SARS-CoV. J Immunol. 2008 Nov 1;181(9):6337-48. doi: 10.4049/jimmunol.181.9.6337. PMID 18941225
- [Background] Bolles M, Deming D, Long K, Agnihothram S, Whitmore A, Ferris M, Funkhouser W, Gralinski L, Totura A, Heise M, Baric RS. A double-inactivated severe acute respiratory syndrome coronavirus vaccine provides incomplete protection in mice and induces increased eosinophilic proinflammatory pulmonary response upon challenge. J Virol. 2011 Dec;85(23):12201-15. doi: 10.1128/JVI.06048-11. Epub 2011 Sep 21. PMID 21937658
- [Background] Tseng CT, Sbrana E, Iwata-Yoshikawa N, Newman PC, Garron T, Atmar RL, Peters CJ, Couch RB. Immunization with SARS coronavirus vaccines leads to pulmonary immunopathology on challenge with the SARS virus. PLoS One. 2012;7(4):e35421. doi: 10.1371/journal.pone.0035421. Epub 2012 Apr 20. PMID 22536382
- [Background] Castilow EM, Olson MR, Varga SM. Understanding respiratory syncytial virus (RSV) vaccine-enhanced disease. Immunol Res. 2007;39(1-3):225-39. doi: 10.1007/s12026-007-0071-6. PMID 17917067
- [Background] Collins PL, Graham BS. Viral and host factors in human respiratory syncytial virus pathogenesis. J Virol. 2008 Mar;82(5):2040-55. doi: 10.1128/JVI.01625-07. Epub 2007 Oct 10. No abstract available. PMID 17928346
- [Background] Deming D, Sheahan T, Heise M, Yount B, Davis N, Sims A, Suthar M, Harkema J, Whitmore A, Pickles R, West A, Donaldson E, Curtis K, Johnston R, Baric R. Vaccine efficacy in senescent mice challenged with recombinant SARS-CoV bearing epidemic and zoonotic spike variants. PLoS Med. 2006 Dec;3(12):e525. doi: 10.1371/journal.pmed.0030525. PMID 17194199
- [Background] Takada A, Kawaoka Y. Antibody-dependent enhancement of viral infection: molecular mechanisms and in vivo implications. Rev Med Virol. 2003 Nov-Dec;13(6):387-98. doi: 10.1002/rmv.405. PMID 14625886
- [Background] Mascola JR, Mathieson BJ, Zack PM, Walker MC, Halstead SB, Burke DS. Summary report: workshop on the potential risks of antibody-dependent enhancement in human HIV vaccine trials. AIDS Res Hum Retroviruses. 1993 Dec;9(12):1175-84. doi: 10.1089/aid.1993.9.1175. PMID 7908211
- [Background] Jaume M, Yip MS, Cheung CY, Leung HL, Li PH, Kien F, Dutry I, Callendret B, Escriou N, Altmeyer R, Nal B, Daeron M, Bruzzone R, Peiris JS. Anti-severe acute respiratory syndrome coronavirus spike antibodies trigger infection of human immune cells via a pH- and cysteine protease-independent FcgammaR pathway. J Virol. 2011 Oct;85(20):10582-97. doi: 10.1128/JVI.00671-11. Epub 2011 Jul 20. PMID 21775467
- [Background] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Background] Wang Q, Zhang L, Kuwahara K, Li L, Liu Z, Li T, Zhu H, Liu J, Xu Y, Xie J, Morioka H, Sakaguchi N, Qin C, Liu G. Immunodominant SARS Coronavirus Epitopes in Humans Elicited both Enhancing and Neutralizing Effects on Infection in Non-human Primates. ACS Infect Dis. 2016 May 13;2(5):361-76. doi: 10.1021/acsinfecdis.6b00006. Epub 2016 Apr 11. PMID 27627203
- [Background] Yip MS, Leung HL, Li PH, Cheung CY, Dutry I, Li D, Daeron M, Bruzzone R, Peiris JS, Jaume M. Antibody-dependent enhancement of SARS coronavirus infection and its role in the pathogenesis of SARS. Hong Kong Med J. 2016 Jun;22(3 Suppl 4):25-31. No abstract available. PMID 27390007
- [Background] Yang ZY, Werner HC, Kong WP, Leung K, Traggiai E, Lanzavecchia A, Nabel GJ. Evasion of antibody neutralization in emerging severe acute respiratory syndrome coronaviruses. Proc Natl Acad Sci U S A. 2005 Jan 18;102(3):797-801. doi: 10.1073/pnas.0409065102. Epub 2005 Jan 10. PMID 15642942
- [Background] Wang SF, Tseng SP, Yen CH, Yang JY, Tsao CH, Shen CW, Chen KH, Liu FT, Liu WT, Chen YM, Huang JC. Antibody-dependent SARS coronavirus infection is mediated by antibodies against spike proteins. Biochem Biophys Res Commun. 2014 Aug 22;451(2):208-14. doi: 10.1016/j.bbrc.2014.07.090. Epub 2014 Jul 26. PMID 25073113
- [Background] Liu L, Wei Q, Lin Q, Fang J, Wang H, Kwok H, Tang H, Nishiura K, Peng J, Tan Z, Wu T, Cheung KW, Chan KH, Alvarez X, Qin C, Lackner A, Perlman S, Yuen KY, Chen Z. Anti-spike IgG causes severe acute lung injury by skewing macrophage responses during acute SARS-CoV infection. JCI Insight. 2019 Feb 21;4(4):e123158. doi: 10.1172/jci.insight.123158. eCollection 2019 Feb 21. PMID 30830861
- [Background] Kam YW, Kien F, Roberts A, Cheung YC, Lamirande EW, Vogel L, Chu SL, Tse J, Guarner J, Zaki SR, Subbarao K, Peiris M, Nal B, Altmeyer R. Antibodies against trimeric S glycoprotein protect hamsters against SARS-CoV challenge despite their capacity to mediate FcgammaRII-dependent entry into B cells in vitro. Vaccine. 2007 Jan 8;25(4):729-40. doi: 10.1016/j.vaccine.2006.08.011. Epub 2006 Aug 22. PMID 17049691
- [Background] Luo F, Liao FL, Wang H, Tang HB, Yang ZQ, Hou W. Evaluation of Antibody-Dependent Enhancement of SARS-CoV Infection in Rhesus Macaques Immunized with an Inactivated SARS-CoV Vaccine. Virol Sin. 2018 Apr;33(2):201-204. doi: 10.1007/s12250-018-0009-2. Epub 2018 Mar 14. No abstract available. PMID 29541941
- [Background] McLellan JS, Chen M, Joyce MG, Sastry M, Stewart-Jones GB, Yang Y, Zhang B, Chen L, Srivatsan S, Zheng A, Zhou T, Graepel KW, Kumar A, Moin S, Boyington JC, Chuang GY, Soto C, Baxa U, Bakker AQ, Spits H, Beaumont T, Zheng Z, Xia N, Ko SY, Todd JP, Rao S, Graham BS, Kwong PD. Structure-based design of a fusion glycoprotein vaccine for respiratory syncytial virus. Science. 2013 Nov 1;342(6158):592-8. doi: 10.1126/science.1243283. PMID 24179220
- [Background] Hadinegoro SR, Arredondo-Garcia JL, Capeding MR, Deseda C, Chotpitayasunondh T, Dietze R, Muhammad Ismail HI, Reynales H, Limkittikul K, Rivera-Medina DM, Tran HN, Bouckenooghe A, Chansinghakul D, Cortes M, Fanouillere K, Forrat R, Frago C, Gailhardou S, Jackson N, Noriega F, Plennevaux E, Wartel TA, Zambrano B, Saville M; CYD-TDV Dengue Vaccine Working Group. Efficacy and Long-Term Safety of a Dengue Vaccine in Regions of Endemic Disease. N Engl J Med. 2015 Sep 24;373(13):1195-206. doi: 10.1056/NEJMoa1506223. Epub 2015 Jul 27. PMID 26214039
- [Background] Kentner AC, Miguelez M, James JS, Bielajew C. Behavioral and physiological effects of a single injection of rat interferon-alpha on male Sprague-Dawley rats: a long-term evaluation. Brain Res. 2006 Jun 20;1095(1):96-106. doi: 10.1016/j.brainres.2006.04.014. Epub 2006 May 18. PMID 16712809
- [Background] Pepini T, Pulichino AM, Carsillo T, Carlson AL, Sari-Sarraf F, Ramsauer K, Debasitis JC, Maruggi G, Otten GR, Geall AJ, Yu D, Ulmer JB, Iavarone C. Induction of an IFN-Mediated Antiviral Response by a Self-Amplifying RNA Vaccine: Implications for Vaccine Design. J Immunol. 2017 May 15;198(10):4012-4024. doi: 10.4049/jimmunol.1601877. Epub 2017 Apr 17. PMID 28416600
- [Background] Geall AJ, Verma A, Otten GR, Shaw CA, Hekele A, Banerjee K, Cu Y, Beard CW, Brito LA, Krucker T, O'Hagan DT, Singh M, Mason PW, Valiante NM, Dormitzer PR, Barnett SW, Rappuoli R, Ulmer JB, Mandl CW. Nonviral delivery of self-amplifying RNA vaccines. Proc Natl Acad Sci U S A. 2012 Sep 4;109(36):14604-9. doi: 10.1073/pnas.1209367109. Epub 2012 Aug 20. PMID 22908294